CLINICAL TRIAL: NCT03823716
Title: Inadvertent Hyperventilation During Intraoperative Care in Neonates
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Kristin Chenault, Clinical Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Other Study IDs: IRB17-00032
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neonatal Disorder
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to evaluate current anesthetic practice in the care of preterm infants and neonates, the investigators will retrospectively review surgical procedures in infants who are less than 60 weeks post-conceptual age in which an arterial cannula was placed intraoperatively or in situ upon arrival in the operating room. They will evaluate the mode of ventilation (pressure or volume-controlled), tidal volume or peak inflating pressure, the level of PEEP, inspired oxygen concentration (FiO2), and respiratory rate used during the procedure to determine the average minute ventilation.

ELIGIBILITY:
Inclusion Criteria:

* neonates (<60 weeks post-conceptual age) undergoing non-cardiac operative procedures in which arterial access is generally present (exploratory laparotomy or thoracotomy)

Exclusion Criteria:

* none

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients seen at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Decreased Partial Pressure of Carbon Dioxide (PaCO2) | During surgical procedure (average of 2-3 hours)
  PaCO2 from arterial blood gas (ABG) ≤ 35

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Chenault, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Chenault K, Wakimoto M, Miller R, Tobias JD. The Incidence and Severity of Hypocarbia in Neonates Undergoing General Anesthesia. Respir Care. 2020 Aug;65(8):1154-1159. doi: 10.4187/respcare.07382. Epub 2020 Mar 17. PMID 32184375